CLINICAL TRIAL: NCT02376179
Title: Endotracheal Tube Intracuff Pressure and Leak Around the Cuff During Retractor Placement for Tonsillectomy and/or Adenoidectomy
Brief Title: Endotracheal Tube Intracuff Pressure and Leak
Status: Completed | Type: Observational
Sponsor: Kris Jatana (Other)
Responsible Party: Sponsor-Investigator, Kris Jatana, ENT Surgeon, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00613
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Otolaryngological Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cuffed ETT: Pediatric patients intubated with a cuffed endotracheal tube for adenotonsillectomy.
  Interventions: Device: Cuffed ETT

INTERVENTIONS:
Device: Cuffed ETT
  Other Names: Kimberly Clark Microcuff ETT

SUMMARY:
We have devised a simple method to continuously measure the endotracheal tube cuff pressure (CP) using an invasive pressure monitoring setup (IPMS), which is used routinely in the operating room to monitor arterial or central venous pressures. We have previously confirmed both in vitro and in vivo (previous IRB approved protocol), a clinically applicable agreement of the IPMS readings with the values obtained from a standard manometer (gold standard). In the current study, we will prospectively evaluate the relationship between the patient's head position and CP in patients undergoing otolaryngological surgery. A secondary outcome measure is the oxygen or nitrous oxygen concentration in the oropharynx.

ELIGIBILITY:
Inclusion Criteria:

* Less than 18 years of age, undergoing otolaryngological surgery with endotracheal intubation.

Exclusion Criteria:

* Patient who is intubated with an uncuffed endotracheal tube.
* Patients who have a limitation for movement of the neck or concerns of the stability of the cervical spine.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Less than 18 years of age, undergoing otolaryngological surgery with endotracheal intubation.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Result] Olsen GH, Krishna SG, Jatana KR, Elmaraghy CA, Ruda JM, Tobias JD. Changes in intracuff pressure of cuffed endotracheal tubes while positioning for adenotonsillectomy in children. Paediatr Anaesth. 2016 May;26(5):500-3. doi: 10.1111/pan.12873. Epub 2016 Mar 9. PMID 26956620

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cuffed ETT
Started | 84
Completed | 84
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cuffed ETT: Pediatric patients intubated with a cuffed endotracheal tube for adenotonsillectomy.
  Cuffed ETT
Arm/Group | Cuffed ETT
Number analyzed (Participants) | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 84
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.7 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 84

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Intracuff Pressure
Description: Changes in the intracuff pressure from baseline of cuffed ETT's after positioning of the patient's head and retractor placement.
Time Frame: during time of surgery
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Cuffed ETT
Number analyzed (Participants) | 84
cmH2O | 3 (7)

ADVERSE EVENTS:
Arm/Group | Cuffed ETT
Serious Adverse Events (participants affected / at risk) | 0/84
Other Adverse Events (participants affected / at risk) | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes